CLINICAL TRIAL: NCT04981626
Title: Interoception in Anorexia Nervosa
Acronym: INT-AN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Santé des Étudiants de France (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00811-40
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-07

CONDITIONS: Anorexia; Anorexia Nervosa; Electrocardiogram; EEG
MeSH Terms: conditions — Anorexia; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: * Females
  * Age : matched for the AN group
  * No present or past eating disorders
  * No past or current psychotic disorders
  * No current substance abuse or dependence.
  * No current psychiatric medication
  Interventions: Other: Clinical and experimental session
- AN group: * Females
  * 16 years ≤ Age ≤ 25 years
  * Diagnostic of AN according to DSM-5 criteria
  * No past or current psychotic disorders
  * No current substance abuse or dependence (excluding tobacco).
  * No current psychiatric medication
  Interventions: Other: Clinical and experimental session

INTERVENTIONS:
Other: Clinical and experimental session — Psychologic profile with standardized interview and scales (see below for details: SCID, BDI, STAI, BPQ, EDE Q, Pictorial Body Image Scale (PBIS) and EDI).
  Measure the stomach-brain synchrony during EEG/EGG resting state, the distribution of voluntary actions across the respiratory phase, and the distribution of saccadic eye movements across the cardiac-cycle.

SUMMARY:
Anorexia nervosa is a serious psychiatric illness whose causes remain poorly understood, and which remains difficult to treat to this day. Many clinical manifestations of this disease can have their origin in abnormalities in the perception of signals coming from inside the body, but this remains to be demonstrated. In recent years, research in healthy subjects has shown how the brain constantly perceives the viscera (heart, lungs, stomach). The examiners will use these new, objective and validated methods to explore how the brain processes information from the viscera (interoception) in anorexic patients. In practice, they will quantify the coupling between the cardiac cycle and involuntary eye movements, as well as between the respiratory cycle and voluntary actions such as pressing a button. Finally, by simultaneously recording the electrical activity of the brain, and that of the stomach, the examiners will measure the coupling between the brain and the stomach. All these measurements, which will be compared between a population of patients and healthy subjects, will make it possible to determine whether anorexic patients have an alteration in the perception of their internal body signals and whether this damage affects several organs.

ELIGIBILITY:
Inclusion Criteria - AN groups:

* Females
* 6 to 25 years old
* Diagnostic of AN according to DSM-5 criteria
* No past or current psychotic disorders
* No current substance abuse or dependence (excluding tobacco).
* No current psychiatric medication

Inclusion Criteria - control groups:

* Females
* Age : matched for the AN group
* No present or past eating disorders
* No past or current psychotic disorders
* No current substance abuse or dependence.
* No current psychiatric medication

Exclusion Criteria for both groups:

* age below 16 years and above 25 years,
* Past or current psychotic disorders,
* Current substance abuse or dependence (excluding tobacco)
* Opposition to participation has been expressed.

In addition, for the control group,

* Subjects with present or past eating disorders or current mental disorders will be excluded.

Ages: 16 Years to 25 Years | Sex: Female
Age Groups: Child, Adult
Study Population: patients with anorexia nervosa (group AN) and healthy control subjects (group C)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
measure brain-stomach interactions using phase-amplitude coupling between the gastric phase and the amplitude of the cortical alpha rhythm. | Experimental session - 10 days maximum after inclusion
  Examiners will directly measure brain-stomach interactions using phase-amplitude coupling between the gastric phase and the amplitude of the cortical alpha rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Solca, Dr, Principal Investigator — ENS
Locations (1):
- ENS, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No